CLINICAL TRIAL: NCT05094349
Title: Influence of Pneumonia on Delayed Cerebral Infarction After Subarachnoid Hemorrhage: a Retrospective Study
Brief Title: Influence of Pneumonia on Delayed Cerebral Ischemia After Subarachnoid Hemorrhage . SAH-CIP (SubArrachnoid Hemorrhage - Cerebral Infarction Pneumonia)
Acronym: SAH-CIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SAH-CIP (29BRC19.0311)
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Subarachnoid Hemorrhage; Pneumonia, Bacterial
Keywords: Subarachnoid hemorrhage; pneumonia; delayed cerebral ischemia; vasospasm; delayed cerebral infarction
MeSH Terms: conditions — Subarachnoid Hemorrhage; Pneumonia, Bacterial; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prognosis of subarachnoid hemorrhage (SAH) is scarce, indeed almost half patients die or become severely disable after SAH. Outcome is related to the severity of the initial bleeding and delayed cerebral infarction (DCI). Infection and more precisely pneumonia have been associated with poor outcome in SAH. However, the interaction between the two pathologic events remains unclear. Therefore, we hypothesized that DCI may be associated to pneumonia in SAH patients. Thus the aim of the study is to analyze the association between delayed cerebral infarction and pneumonia in patients with SAH.

Retrospective, observational, monocentric cohort study, including patient admitted in Neurosurgical Intensive Care Unit or Surgical Intensive Care Unit in the University Hospital of Brest (France) for non-traumatic SAH. Primary outcome is diagnosis of DCI on CT scan or MRI 3 months after SAH. Multivariate analysis is used to identify factors independently associated with DCI.

We plan to include between 200 and 250 patients in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* admitted in ICU in Brest University Hospital
* for non traumatic subarachnoid hemorrhage
* between july 2015 and december 2018

Exclusion Criteria:

* continuation of care out of Brest University Hospital after initial ICU stay
* refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient admitted to ICU for subarachnoid hemorrhage (SAH). in our institution every patient diagnosed with non traumatic SAH are admitted for at least 24 hours in ICU.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
delayed cerebral infarction | 3 months from subarachnoid hemorrhage
  infarction on CT or MRI not related to initial bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 2 years and ending five years following the end of study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.